CLINICAL TRIAL: NCT06853678
Title: Selinexor Combined With Nab-paclitaxel and Adebrelimab as Second-line Treatment for ES-SCLC：A Prospective, Single-center, Single-arm Clinical Study
Brief Title: Second-line Immunotherapy for ES-SCLC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ES-SCLC-001
Record Dates: First submitted 2025-02-25; First posted 2025-03-03 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Extensive Stage Small Cell Lung Cancer (ES-SCLC)
MeSH Terms: interventions — selinexor; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental): Immunotherapy combined with chemotherapy
  Interventions: Drug: Adebrelimab; Drug: Selinexor; Drug: Nab-paclitaxel

INTERVENTIONS:
Drug: Adebrelimab — 1200mg,d1,iv,q3w
Drug: Selinexor — 40mg,twice weekly,d1, d3,oral,q3w
Drug: Nab-paclitaxel — 100mg/m2,d1,d8,d15,iv,q3w

SUMMARY:
At present, the first-line standard treatment for patients with extensive-stage small cell lung cancer (ES-SCLC) is immunotherapy combined with chemotherapy. For patients who relapse within 6 months after first-line chemotherapy, conventionally recommended chemotherapy drugs include topotecan, irinotecan, gemcitabine, paclitaxel or vinorelbine, etc., but due to limited benefits to patients, patients are also recommended to participate in relevant clinical studies. New treatment methods are constantly being explored in second-line treatment, including fluzoparib combined with adebelimumab. The current status of second-line treatment is still worrying.

Selinexor is a class of nuclear export selective inhibitors (SINEs) for the export protein receptor XPO1. PO1 promotes the transport of mRNA and cargo proteins, including tumor suppressor proteins (TSPs), hormone receptors (GRs), and immune response regulators. Selinexor covalently binds to the XPO1 protein, blocking the export of TSPs and GRs and accumulating them in the nucleus, preventing the translation of oncoprotein mRNA, stopping the cell cycle process, and initiating apoptosis. Multiple in vitro and in vivo studies have verified that selinexor combined with chemotherapy/radiotherapy/targeted therapy exhibits significant anti-tumor activity.

This study plans to use selinexor combined with adebrelimab and albumin-paclitaxel as a second-line treatment for ES-SCLC to explore the efficacy and safety of this regimen.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old, male or female;
* ECOG PS score 0-1 points;
* Expected survival period is not less than 12 weeks;
* Patients with pathologically (histologically or cytologically) confirmed small cell lung cancer (according to the 2015 classification of the World Health Organization);
* Patients with extensive stage small cell lung cancer confirmed by imaging (staging according to the eighth edition of TNM staging);
* With measurable lesions (according to RECIST 1.1 standards, the long diameter of the tumor lesion on CT scan is ≥ 10mm);
* Need to have failed standard first-line treatment before enrollment;
* Agree to collect tumor histological specimens required for this study and use them in related research;
* Main organ function is normal, without severe abnormal blood, heart, lung, liver, kidney function and immunodeficiency diseases.
* Female subjects of childbearing potential must undergo a serum or urine pregnancy test within 72 hours before starting the trial drug, and the result must be negative, and they must be willing to use a medically approved high-efficiency contraceptive method (such as intrauterine contraceptive device, contraceptive pills or condoms) during the study and within 90 days after the last administration of the trial drug; male subjects whose partners are female subjects of childbearing potential should be surgically sterilized or agree to use effective contraceptive methods during the study and within 90 days after the last administration of the trial drug.
* Subjects voluntarily join this study and sign the Informed Consent Form (ICF), have good compliance, and can follow up the efficacy and adverse reactions as required by the protocol

Exclusion Criteria:

* Any active autoimmune disease or history of autoimmune disease with expected recurrence (including but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism [subjects who can be controlled only by hormone replacement therapy can be included]; subjects with skin diseases that do not require systemic treatment such as vitiligo, psoriasis, alopecia, type I diabetes or asthma that has been completely relieved in childhood and does not require any intervention in adulthood can be included; asthma patients who require bronchodilators for medical intervention are not included);
* Suffering from congenital or acquired immune deficiency, such as human immunodeficiency virus (HIV) infection, untreated active hepatitis B (HBsAg positive or HBV DNA ≥ 500 IU/ml and abnormal liver function), hepatitis C (positive hepatitis C antibody, and HCV-RNA is higher than the detection limit of the analytical method and liver function is abnormal) or co-infection with hepatitis B and hepatitis C;
* Subjects who need systemic treatment with corticosteroids (>10 mg/day of prednisone or equivalent dose of similar hormones) or other immunosuppressants within 14 days before the first use of the trial drug;
* Subjects who received live attenuated vaccines within 4 weeks before the first dose or planned to receive them during the study;
* Subjects who have previously or are currently using any other anti-tumor treatment for SCLC;
* Subjects who have suffered from malignant tumors other than SCLC in the past 5 years, excluding fully treated cervical carcinoma in situ, basal cell or squamous cell skin cancer, localized prostate cancer after radical surgery, and ductal carcinoma in situ after radical surgery;
* Evidence of past or current pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonia, drug-induced pneumonia, and severe lung function impairment;
* Suffering from grade II or above myocardial ischemia or myocardial infarction, and poorly controlled arrhythmias (including QTc interval ≥450ms for men and ≥470ms for women). According to NYHA standards, patients with grade III-IV heart failure, or left ventricular ejection fraction (LVEF) <50% indicated by cardiac ultrasound examination, had the following conditions within 6 months before entering the study: myocardial infarction, severe/unstable angina, NYHA grade 2 or above heart failure, and clinically significant supraventricular or ventricular arrhythmias requiring clinical intervention;
* Urinalysis indicated urine protein ≥ (++), or 24-hour urine protein ≥ 1.0 g;
* Patients with thrombotic diseases requiring long-term anticoagulation therapy with warfarin or heparin, or requiring long-term antiplatelet therapy (aspirin ≥ 300 mg/day or clopidogrel ≥ 75 mg/day);
* Systemic antibiotics used for ≥7 days within 4 weeks before the first dose, or unexplained fever >38.5℃ during the screening period/before the first dose (fever caused by tumors can be included in the study as determined by the investigator);
* Known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation;
* Pregnant or lactating women; patients of fertile potential who are unwilling or unable to take effective contraceptive measures;
* Known allergic reactions, hypersensitivity reactions, or intolerance to carrelizumab and other monoclonal antibodies, pemetrexed, albumin-paclitaxel, prophylactic medications, or their excipients;
* Any condition that the investigator believes may harm the subject or cause the subject to be unable to meet or perform the study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-02-28 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival，PFS | 24months
  From randomization to tumor progression (of any kind) or death (from any cause).

SECONDARY OUTCOMES:
Objective response rate，ORR | 24months
  The proportion of patients whose tumor volume has decreased to a predetermined value and was defined as the percentage of patients with CR and PR.
Disease control rate, DCR | 24months
  DCR was defined based on the cumulative objective response and stabilization rates (CR+PR+SD).
Overall survival，OS | 24months
  Time from randomization to death from any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No